CLINICAL TRIAL: NCT03655223
Title: Early Check: A Collaborative Innovation to Facilitate Pre-Symptomatic Clinical Trials in Newborns
Brief Title: Early Check: Expanded Screening in Newborns
Status: Enrolling by invitation | Type: Observational
Sponsor: RTI International (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); The John Merck Fund (Unknown); Duke University (Other); Wake Forest University (Other); North Carolina Department of Health and Human Services (Other Government); National Center for Advancing Translational Sciences (NCATS) (NIH); Cure SMA (Other); The National Fragile X Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Asuragen, Inc. (Unknown); Sarepta Therapeutics, Inc. (Industry); Muscular Dystrophy Association (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); Juvenile Diabetes Research Foundation (Other); Janssen Pharmaceuticals (Industry); GeneDx (Unknown); Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-0009; HHSN27500003 (Other Grant/Funding Number: Eunice Kennedy Shriver National Institute of Child Health and Human Development)
Record Dates: First submitted 2018-08-16; First posted 2018-08-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-12

CONDITIONS: Spinal Muscular Atrophy; Fragile X Syndrome; Fragile X - Premutation; Duchenne Muscular Dystrophy; Hyperinsulinemic Hypoglycemia, Familial 1; Diabetes Mellitus; Adrenoleukodystrophy, Neonatal; Medium-chain Acyl-CoA Dehydrogenase Deficiency; Very Long Chain Acyl Coa Dehydrogenase Deficiency; Beta-ketothiolase Deficiency; Severe Combined Immunodeficiency Due to Adenosine Deaminase Deficiency; Primary Hyperoxaluria Type 1; Congenital Bile Acid Synthesis Defect Type 2; Pyridoxine-Dependent Epilepsy; Hereditary Fructose Intolerance; Hypophosphatasia; Hyperargininemia; Mucopolysaccharidosis Type 6; Argininosuccinic Aciduria; Citrullinemia, Type I; Wilson Disease; Maple Syrup Urine Disease, Type 1A; Maple Syrup Urine Disease, Type 1B; Biotinidase Deficiency; Neonatal Severe Primary Hyperparathyroidism; Intrinsic Factor Deficiency; Usher Syndrome Type 1D/F Digenic (Diagnosis); Cystic Fibrosis; Stickler Syndrome Type 2; Stickler Syndrome Type 1; Alport Syndrome, Autosomal Recessive; Alport Syndrome, X-Linked; Carbamoyl Phosphate Synthetase I Deficiency Disease; Carnitine Palmitoyl Transferase 1A Deficiency; Carnitine Palmitoyltransferase II Deficiency; Cystinosis; Chronic Granulomatous Disease; Cerebrotendinous Xanthomatoses; Maple Syrup Urine Disease, Type 2; Severe Combined Immunodeficiency Due to DCLRE1C Deficiency; Thyroid Dyshormonogenesis 6; Thyroid Dyshormonogenesis 5; Supravalvar Aortic Stenosis; Factor X Deficiency; Hemophilia A; Hemophilia B; Tyrosinemia, Type I; Fructose 1,6 Bisphosphatase Deficiency; Glycogen Storage Disease Type I; G6PD Deficiency; Glycogen Storage Disease II; Galactokinase Deficiency; Mucopolysaccharidosis Type IV A; Galactosemias; Guanidinoacetate Methyltransferase Deficiency; Agat Deficiency; Glutaryl-CoA Dehydrogenase Deficiency; Gtp Cyclohydrolase I Deficiency; Hyperinsulinism-Hyperammonemia Syndrome; Primary Hyperoxaluria Type 2; 3-Hydroxyacyl-CoA Dehydrogenase Deficiency; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; Mitochondrial Trifunctional Protein Deficiency; Sickle Cell Disease; Beta-Thalassemia; Holocarboxylase Synthetase Deficiency; 3-Hydroxy-3-Methylglutaric Aciduria; Primary Hyperoxaluria Type 3; Hermansky-Pudlak Syndrome 1; Hermansky-Pudlak Syndrome 4; Apparent Mineralocorticoid Excess; HSDB; CBAS1; Mucopolysaccharidosis Type 2; Mucopolysaccharidosis Type 1; Severe Combined Immunodeficiency, X Linked; Severe Combined Immunodeficiency Due to IL-7Ralpha Deficiency; Diabetes Mellitus, Permanent Neonatal; Isovaleric Acidemia; Severe Combined Immunodeficiency T-Cell Negative B-Cell Positive Due to Janus Kinase-3 Deficiency (Disorder); Jervell and Lange-Nielsen Syndrome 2; Hyperinsulinemic Hypoglycemia, Familial, 2; Diabetes Mellitus, Permanent Neonatal, With Neurologic Features; Jervell and Lange-Nielsen Syndrome 1; Lysosomal Acid Lipase Deficiency; CblF; 3-Methylcrotonyl CoA Carboxylase 1 Deficiency; 3-Methylcrotonyl CoA Carboxylase 2 Deficiency; Waardenburg Syndrome Type 2A; Methylmalonic Aciduria cblA Type; Methylmalonic Aciduria cblB Type; Methylmalonic Aciduria and Homocystinuria Type cblC; MAHCD; Methylmalonic Aciduria Due to Methylmalonyl-CoA Mutase Deficiency; Congenital Disorder of Glycosylation Type 1B; Mthfr Deficiency; Methylcobalamin Deficiency Type Cbl G (Disorder); Methylcobalamin Deficiency Type cblE; Usher Syndrome, Type 1B; N-acetylglutamate Synthase Deficiency; Ornithine Transcarbamylase Deficiency; Phenylketonurias; Waardenburg Syndrome Type 1; Congenital Hypothyroidism; Propionic Acidemia; Usher Syndrome, Type 1F; Pancreatic Agenesis 1; Hereditary Hypophosphatemic Rickets; Glycogen Storage Disease IXB; Glycogen Storage Disease IXC; MOWS; Epilepsy, Early-Onset, Vitamin B6-Dependent; Pyridoxal Phosphate-Responsive Seizures; Pituitary Hormone Deficiency, Combined, 1; Ptsd; Dihydropteridine Reductase Deficiency; Severe Combined Immunodeficiency Due to RAG1 Deficiency; Severe Combined Immunodeficiency Due to RAG2 Deficiency; Retinoblastoma; Multiple Endocrine Neoplasia Type 2B; Pseudohypoaldosteronism, Type I; Liddle Syndrome; Biotin-Responsive Basal Ganglia Disease; SCD; DIAR1; GSD1C; Acrodermatitis Enteropathica; Thyroid Dyshormonogenesis 1; Riboflavin Transporter Deficiency; Waardenburg Syndrome, Type 2E; SRD; Congenital Lipoid Adrenal Hyperplasia Due to STAR Deficiency; Barth Syndrome; Adrenocorticotropic Hormone Deficiency; Transcobalamin II Deficiency; Thyroid Dyshormonogenesis 3; Segawa Syndrome, Autosomal Recessive; Autosomal Recessive Nonsyndromic Hearing Loss; Thyroid Dyshormonogenesis 2A; Congenital Isolated Thyroid Stimulating Hormone Deficiency; Hypothyroidism Due to TSH Receptor Mutations; Usher Syndrome Type 1C; Usher Syndrome Type 1G (Diagnosis); Von Willebrand Disease, Type 3; Combined Immunodeficiency Due to ZAP70 Deficiency; Adenine Phosphoribosyltransferase Deficiency; Metachromatic Leukodystrophy; Canavan Disease; Menkes Disease; Carbonic Anhydrase VA Deficiency; Developmental and Epileptic Encephalopathy 2; 17 Alpha-Hydroxylase Deficiency; Smith-Lemli-Opitz Syndrome; Krabbe Disease; Glutathione Synthetase Deficiency; Mucopolysaccharidosis Type 7; Rett Syndrome; Molybdenum Cofactor Deficiency, Type A; Niemann-Pick Disease, Type C1; Niemann-Pick Disease Type C2; Ornithine Aminotransferase Deficiency; 3-Phosphoglycerate Dehydrogenase Deficiency; Leber Congenital Amaurosis 2; Dravet Syndrome; Mucopolysaccharidosis Type 3 A; Ornithine Translocase Deficiency; Carnitine-acylcarnitine Translocase Deficiency; Glucose Transporter Type 1 Deficiency Syndrome; Creatine Transporter Deficiency; Niemann-Pick Disease Type A; Pitt Hopkins Syndrome; Tuberous Sclerosis 1; Tuberous Sclerosis 2; Ataxia With Isolated Vitamin E Deficiency; Angelman Syndrome; Prader-Willi Syndrome; Homocystinuria; Permanent Neonatal Diabetes Mellitus; Transient Neonatal Diabetes Mellitus; Factor VII Deficiency; Glycogen Storage Disease Type IXA1; Glycogen Storage Disease, Type IXA2; Glycogen Storage Disease IC; Glycogen Storage Disease Type IB; Central Hypoventilation Syndrome With or Without Hirschsprung Disease
Keywords: Newborn Screening; Rare Disorders; Genetic Counseling; Families; Development; Risk; Genetic Sequencing
MeSH Terms: conditions — Muscular Atrophy, Spinal; Fragile X Syndrome; Muscular Dystrophy, Duchenne; Congenital Hyperinsulinism; Diabetes Mellitus; Peroxisomal Disorders; Medium chain acyl CoA dehydrogenase deficiency; VLCAD deficiency; Beta ketothiolase deficiency; Severe combined immunodeficiency due to adenosine deaminase deficiency; Primary hyperoxaluria type 1; Bile acid synthesis defect, congenital, 2; Pyridoxine-dependent epilepsy; Fructose Intolerance; Hypophosphatasia; Hyperargininemia; Mucopolysaccharidosis VI; Argininosuccinic Aciduria; Citrullinemia; Hepatolenticular Degeneration; Maple syrup urine disease, type 1A; Maple syrup urine disease, type 1B; Biotinidase Deficiency; Hyperparathyroidism, Neonatal Severe Primary; Intrinsic Factor Deficiency; Disease; Cystic Fibrosis; Stickler syndrome, type 2; Stickler syndrome, type 1; Nephritis, Hereditary; Carbamoyl-Phosphate Synthase I Deficiency Disease; Carnitine palmitoyl transferase 1A deficiency; Carnitine palmitoyl transferase 2 deficiency; Cystinosis; Granulomatous Disease, Chronic; Xanthomatosis, Cerebrotendinous; Maple syrup urine disease, type 2; Thyroid Dyshormonogenesis 6; Thyroid Dyshormonogenesis 5; Aortic Stenosis, Supravalvular; Factor X Deficiency; Hemophilia A; Hemophilia B; Tyrosinemias; Fructose-1,6-Diphosphatase Deficiency; Glycogen Storage Disease Type I; Glucosephosphate Dehydrogenase Deficiency; Glycogen Storage Disease Type II; Galactosemias; Mucopolysaccharidosis IV; Guanidinoacetate methyltransferase deficiency; Arginine-Glycine Amidinotransferase Deficiency; Glutaric Acidemia I; Hyperphenylalaninemia, BH4-Deficient, B; Hyperinsulinemic hypoglycemia, familial, 6; Primary hyperoxaluria type 2; 3-Hydroxyacyl-CoA Dehydrogenase Deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Anemia, Sickle Cell; beta-Thalassemia; Holocarboxylase Synthetase Deficiency; 3-Hydroxy-3-Methylglutaryl-CoA Lyase Deficiency; Hermanski-Pudlak Syndrome; Mineralocorticoid Excess Syndrome, Apparent; Mucopolysaccharidosis II; Mucopolysaccharidosis I; X-Linked Combined Immunodeficiency Diseases; Diabetes Mellitus, Permanent Neonatal; Acidemia, isovaleric; Jervell And Lange-Nielsen Syndrome 2; Diabetes Mellitus, Permanent Neonatal, With Neurologic Features; Jervell-Lange Nielsen Syndrome; Wolman Disease; 3-methylcrotonyl CoA carboxylase 1 deficiency; 3-methylcrotonyl CoA carboxylase 2 deficiency; Waardenburg syndrome type 2A; Methylmalonic aciduria cblA type; Methylmalonic aciduria cblB type; Methylmalonic acidemia with homocystinuria; Methylmalonic Aciduria due to Methylmalonyl-CoA Mutase Deficiency; Congenital disorder of glycosylation type 1B; Methylenetetrahydrofolate reductase deficiency; Homocystinuria-Megaloblastic Anemia due to Defect in Cobalamin Metabolism, CblE Complementation Type; Usher syndrome, type 1B; N-acetyl glutamate synthetase deficiency; Ornithine Carbamoyltransferase Deficiency Disease; Phenylketonurias; Waardenburg Syndrome; Congenital Hypothyroidism; Propionic Acidemia; Usher syndrome, type 1F; Maturity-Onset Diabetes of the Young, Type 4; Familial Hypophosphatemic Rickets; Glycogen Storage Disease IXB; Glycogen Storage Disease IXC; Epilepsy; Pyridoxamine 5-Prime-Phosphate Oxidase Deficiency; Pituitary Hormone Deficiency, Combined, 1; Stress Disorders, Post-Traumatic; Retinoblastoma; Multiple Endocrine Neoplasia Type 2b; Pseudohypoaldosteronism; Liddle Syndrome; Basal ganglia disease, biotin-responsive; Acrodermatitis enteropathica; Thyroid Dyshormonogenesis 1; Brown-Vialetto-Van Laere syndrome; Waardenburg syndrome type 2; Barth Syndrome; Adrenocorticotropic hormone deficiency; Thyroid Dyshormonogenesis 3; Segawa syndrome, autosomal recessive; Thyroid Dyshormonogenesis 2A; Usher syndrome, type 1C; von Willebrand Disease, Type 3; Adenine phosphoribosyltransferase deficiency; Leukodystrophy, Metachromatic; Canavan Disease; Menkes Kinky Hair Syndrome; Epilepsies, Myoclonic; Adrenal hyperplasia, congenital, type 5; Smith-Lemli-Opitz Syndrome; Leukodystrophy, Globoid Cell; Glutathione synthetase deficiency; Mucopolysaccharidosis VII; Rett Syndrome; Molybdenum Cofactor Deficiency, Complementation Group A; Niemann-Pick Disease, Type C; Niemann-Pick disease, type C2; Gyrate Atrophy; Amaurosis congenita of Leber, type 2; Mucopolysaccharidosis III; HHH syndrome; Carnitine-Acylcarnitine Translocase Deficiency; Glut1 Deficiency Syndrome; Creatine deficiency, X-linked; Niemann-Pick Disease, Type A; Pitt-Hopkins syndrome; Tuberous Sclerosis 1; Tuberous Sclerosis 2; Ataxia with vitamin E deficiency; Angelman Syndrome; Prader-Willi Syndrome; Homocystinuria; Factor VII Deficiency; Glycogen Storage Disease, Type IXA2; Glycogen Storage Disease IC; Glycogen Storage Disease IB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any biological specimens collected as part of the study will be incinerated at the conclusion of the study. Specimens utilized during the study that were collected as part of routine State newborn screening or diagnostic confirmatory testing, will be retained by the North Carolina State Laboratory of Public Health (NCSLPH),University of North Carolina at Chapel Hill (UNC), Invitae, and LabCorps in accordance with institute record retention policies and protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Newborn infants born in North Carolina: All newborn infants in North Carolina will have the opportunity to participate in Early Check. Those who screen positive for the conditions identified in the study will be subject to confirmatory testing.
  Interventions: Diagnostic Test: Confirmatory Testing
- Birthing Mothers in North Carolina: All birthing mothers in North Carolina will have the opportunity to participate in Early Check.

INTERVENTIONS:
Diagnostic Test: Confirmatory Testing — If a newborn's screening test is positive, an experienced genetic counselor will contact the infant's mother by phone to explain the positive screening result and arrange for confirmatory testing and a follow-up appointment. If the confirmatory test is positive, then the child receives a diagnosis of the disease. Children identified with a disorder are referred for treatment, their parents receive information and counseling on what a positive diagnosis means for their child, and they are offered participation in follow-up and registry activities for the disorder.
  Groups: Newborn infants born in North Carolina

SUMMARY:
Early Check provides voluntary screening of newborns for a selected panel of conditions. The study has three main objectives: 1) develop and implement an approach to identify affected infants, 2) address the impact on infants and families who screen positive, and 3) evaluate the Early Check program. The Early Check screening will lead to earlier identification of newborns with rare health conditions in addition to providing important data on the implementation of this model program. Early diagnosis may result in health and development benefits for the newborns. Infants who have newborn screening in North Carolina will be eligible to participate, equating to over 120,000 eligible infants a year. Over 95% of participants are expected to screen negative. Newborns who screen positive and their parents are invited to additional research activities and services. Parents can enroll eligible newborns on the Early Check electronic Research Portal. Screening tests are conducted on residual blood from existing newborn screening dried blood spots. Confirmatory testing is provided free-of-charge for infants who screen positive, and carrier testing is provided to mothers of infants with fragile X. Affected newborns have a physical and developmental evaluation. Their parents have genetic counseling and are invited to participate in surveys and interviews. Ongoing evaluation of the program includes additional parent interviews.

DETAILED DESCRIPTION:
"Background" Newborn screening (NBS) is a state-based public health program that screens babies for a panel of over 30 conditions. It is estimated that about 12,500 newborns each year in the United States are identified with one of the conditions screened in NBS, with each child receiving the benefit of early treatment. For inclusion in newborn screening there must be evidence that pre-symptomatic treatment is more effective than treatment after clinical presentation. Most conditions proposed for newborn screening are rare, however, and researchers have difficulty identifying sufficient numbers of babies to test the benefits of pre-symptomatic identification and treatment. This lack of data is central to challenges that the U.S. Department of Health and Human Services Advisory Committee on Heritable Disorders in Newborns and Children (ACHDNC) faces when making federal recommendations to states on which conditions should be included in newborn screening programs. ACHDNC is often asked to consider conditions for inclusion in newborn screening for which there is limited evidence of the natural history, prevalence, and especially about the benefit of early treatment.

"Rationale" That evidence gap, especially in the rare disease context, makes it important to develop and test a system to efficiently generate high-quality data about conditions that have the potential to be candidates for state newborn screening. The Early Check program will address this gap through screening newborns for a carefully selected panel of conditions, offered under a research protocol with biological maternal permission, except in cases where there is a transfer or loss of custody. In cases with a transfer/loss of custody, a legal guardian can grant permission for the infant to join Early Check. Early Check will identify pre-symptomatic infants with rare disorders, accelerate the acquisition of data on the early natural history of rare disorders, and demonstrate the feasibility of a statewide program to offer voluntary opt-in newborn screening for a panel of conditions not currently included in states' standard newborn screening. Further, Early Check will facilitate the public health 'on-boarding' of conditions that are ultimately recommended for state newborn screening programs.

The initial panel of conditions screened in the Early Check program will change over the course of the study. Previously screened conditions have included spinal muscular dystrophy (SMA), fragile X syndrome (FXS), and Duchenne muscular dystrophy (DMD) and related neuromuscular conditions that result in increased levels of creatine kinase (CK-MM). SMA has an approved treatment, nusinersen, which has been demonstrated to improve outcomes in infants with infantile-onset SMA. In addition, infants with a shorter disease duration compared to a longer disease duration had improved outcomes after the start of treatment with nusinersen, suggesting that earlier identification of SMA would benefit affected infants. There is also an approved gene therapy, Zolgensma, for SMA. FXS does not have an approved treatment, although there is evidence that early behavioral intervention services may improve outcomes. Given that the diagnosis of FXS is made on average after the child is three years old, early identification through the screening of newborns may provide benefit to the child. These conditions are rare; SMA has an estimated incidence of 1 in ~10,000, DMD has an estimated incidence of 1 in 4000-5000 males, and FXS has an estimated incidence of 1 in ~4,000 males and 1 in ~4,000-6,000 females. We also completed a sub-study with a secondary permission process that offers mothers the choice to obtain additional data about the gene that causes FXS: specifically, whether the infant has a premutation in the gene, which has an uncertain impact on the infant's learning and development. This uncertainty is the reason why premutation results are offered separately under a sub-study. DMD causes progressive inflammation, fibrosis, and muscle fiber degradation, and weakness. DMD has traditionally been treated with physical therapy, corticosteroids, and ACE inhibitors to delay the progression of skeletal muscle and cardiac damage. In 2016, the FDA approved Eteplirsen (Exondys, 51) a promising treatment for a subset of patients with DMD. In 2017 the FDA approved Emflaza, a corticosteroid also known as deflazacort. In 2019 the FDA approved Vyondys 53 and in 2020 the FDA approved Viltepso for mutations amenable to exon 53 skipping. Early diagnosis allows for treatments that might work best if used presymptomatically.

The current screening panel includes 182 genes for rare conditions that are highly actionable by age 2. An optional secondary panel includes 32 genes that are less actionable, or for which there are treatments under trial, with an additional optional third panel that screens for genetic risk for Type 1 Diabetes.

For a wide range of rare disorders there is evidence that a delayed diagnosis (i.e., the frequently-described diagnostic odyssey as parents search for a diagnosis) can have negative health outcomes on children who miss out on treatments or interventions and on families who experience negative psychosocial impact

In the future, Early Check will continue to integrate new conditions to the screening platform as science advances and funding is secured, and conditions may be removed from the screening platform as associated research questions are answered and/or conditions achieve inclusion in state newborn screening programs (as was the case with SMA and FXS).

The overall research question is whether Early Check is an effective onboarding program to inform newborn screening policy decision-making.

Early Check will also provide the infrastructure to facilitate translational research studies and clinical trials. A dilemma in research in rare diseases is a lack of sufficient numbers of presymptomatic patients. New treatments are being developed for rare diseases at a rapid pace. Presymptomatic treatment often has the best potential for effective treatment. Currently, early identification and intervention is based on the prenatal or early diagnosis of a sibling of a patient with known disease, which greatly limits the numbers of presymptomatic patients available for trials. Newborn screening has the greatest potential to identify presymptomatic infants. Ultimately the research program should more rapidly advance understanding of diseases and treatments, reducing the length of time for appropriate conditions to be added to the recommended panel for inclusion in state newborn screening programs, and provide early identification of affected newborns.

Overall, this project will provide important information about the success of Early Check to feasibly and acceptably implement a large scale, electronically-mediated research approach to accurately identify affected infants. Results of the research activities and the ongoing quality assessment will be used to inform the most efficient and judicious translation of expanded newborn screening into public health in ways that maximize benefit and minimize potential risk of harm to children and families.

ELIGIBILITY:
Inclusion Criteria:

* Newborn has newborn screening in North Carolina
* Newborn lives in North Carolina or South Carolina
* Newborn is less than 31 days old
* Person giving consent must have legal custody of the newborn. When the mother retains custody, they must be the person to give consent.
* Person giving consent must be able to interact with the online permission portal (available in English and Spanish) and give permission online

Exclusion Criteria:

* A newborn screening (NBS) sample is unavailable for the newborn
* Insufficient NBS sample remains to conduct the screening

Ages: 1 Day to 31 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns born in North or South Carolina who are less than 31 days old
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence Rates: Number of newborns who screen positive comparative to the whole sample | Every 6 months for approximately three years
  Incidence rates of infants who screen positive for conditions on the Early Check panel.

SECONDARY OUTCOMES:
Impact of Screening: Semi-structured parent interviews. | Measured within 6 months of participant screening results
  Each project year, we will recruit mothers whose newborns screen negative and mothers whose newborns screen positive to participate in an approximately 30-minute, semi-structured telephone interview about their perceptions of Early Check and the impact of screening results.

CONTACTS AND LOCATIONS:
Overall Officials: Don Bailey, PhD, Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finkel, Mercuri, Darras, Kuntz, Kirschner et al, 2017
- [Background] Birnkrant, et al, 2018
- [Background] Winarni, Schneider, Borodyanskara, & Hagerman, 2012
- [Background] Bailey, Raspa, Bishop & Holiday, 2009
- [Derived] Gehtland LM, Paquin RS, Andrews SM, Lee AM, Gwaltney A, Duparc M, Pfaff ER, Bailey DB Jr. Using a Patient Portal to Increase Enrollment in a Newborn Screening Research Study: Observational Study. JMIR Pediatr Parent. 2022 Feb 10;5(1):e30941. doi: 10.2196/30941. PMID 35142618
- [Derived] Bailey DB Jr, Gehtland LM, Lewis MA, Peay H, Raspa M, Shone SM, Taylor JL, Wheeler AC, Cotten M, King NMP, Powell CM, Biesecker B, Bishop CE, Boyea BL, Duparc M, Harper BA, Kemper AR, Lee SN, Moultrie R, Okoniewski KC, Paquin RS, Pettit D, Porter KA, Zimmerman SJ. Early Check: translational science at the intersection of public health and newborn screening. BMC Pediatr. 2019 Jul 17;19(1):238. doi: 10.1186/s12887-019-1606-4. PMID 31315600